CLINICAL TRIAL: NCT01143922
Title: Role of Intraoperative Ultrasound in Gastrointestinal (GI) Malignancies
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: All India Institute of Medical Sciences (Other)
Responsible Party: Gaurav N Chaubal, AIIMS
Other Study IDs: IOUS
Record Dates: First submitted 2010-06-14; First posted 2010-06-15 (Estimated); Last update posted 2010-06-15 (Estimated); Status verified 2010-01

CONDITIONS: Ultrasonography; Gastrointestinal Disease; Malignancy
Keywords: Intraoperative ultrasound; GI tract malignancies; modality; ultrasound; staging modality
MeSH Terms: conditions — Gastrointestinal Diseases; Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Patients with gastrointestinal tract malignancies: All patients with GI tract malignancies undergoing surgery will be subjected to intraoperative ultrasound

SUMMARY:
Currently available investigating modalities like CT scans, MRI etc although have a high accuracy in staging of gastrointestinal(GI) tract malignancies, are not correct in all cases . The aim of this study is to assess the role of intraoperative ultrasound as a modality to increase the staging accuracy of GI tract malignancies

ELIGIBILITY:
Inclusion Criteria:

* Patients with GI tract malignancies

Exclusion Criteria:

* Patients who refuse consent

Ages: 10 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: All patients with GI tract malignancies undergoing surgery
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2009-08

CONTACTS AND LOCATIONS:
Locations (1):
- AIIMS, New Delhi, National Capital Territory of Delhi, India